CLINICAL TRIAL: NCT03050931
Title: Imaging Stroke, Epilepsy and Evoked Potentials in the Brain Using Electrical Impedance Tomography
Brief Title: Electrical Impedance Tomography of Epilepsy
Status: Active, not recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 14/0861a
Record Dates: First submitted 2017-02-08; First posted 2017-02-13 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Epilepsy
Keywords: Electrical Impedance Tomography; EIT; Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Epilepsy with intracranial electrodes: Electrical Impedance Tomography with depth electrodes or intracranial electrode mats
  Interventions: Device: Electrical Impedance Tomography
- Epilepsy with scalp electrodes: Electrical Impedance Tomography with scalp electrodes
  Interventions: Device: Electrical Impedance Tomography

INTERVENTIONS:
Device: Electrical Impedance Tomography — EIT comprises of a box of electronics similar in size to a video recorder, laptop computer and leads which link typically to 16 or 32 external ECG-like electrodes placed around the subject. Images are generated by applying tiny electrical signals through some electrodes and recording the resulting signals at others. The signals applied are completely safe, within established British and EU safety limits and cannot be felt. For intracranial electrode studies, the EIT systems will be linked to the existing EEG video recording systems and EIT will be recorded at the same time using some or all of the available intracranial electrodes.
  Other Names: EIT

SUMMARY:
The purpose of this study is to determine if Electrical Impedance Tomography (EIT) can produce reproducible and accurate images in people with epilepsy compared to existing standards such as MRI, CT or EEG.

Electrical Impedance Tomography is a relatively new medical imaging method, which has the potential to provide novel images of brain function. It is fast, portable, safe and inexpensive, but currently has a relatively poor spatial resolution. It produces images of the internal electrical impedance of a subject with epilepsy using rings of ECG like electrodes on the skin, intracranial electrode mats or deep electrodes implemented surgically as part of clinical assessment. EIT recording will take place in parallel with the routine recording on the ward. Following completion of the recording, the EIT images will subsequently be analysed and compared to other imaging data for accuracy.

DETAILED DESCRIPTION:
Electrical Impedance Tomography (EIT) is a novel medical imaging method in which tomographic images are rapidly produced using electrodes placed around the body. The principal applicant's group has demonstrated that EIT can rapidly image functional brain activity in stroke, epilepsy and normal activity in animal models and has developed instrumentation and image reconstruction algorithms which work well in head-shaped tanks.

The principal aim of this research is to optimise and assess accuracy of Electrical Impedance Tomography (EIT) using scalp electrodes, intracranial electrode mats or deep electrodes in imaging epilepsy in human participants. If successful, EIT has the potential to provide a new portable imaging unit. It could be used with scalp electrodes and enable imaging of the onset and propagation of seizures in 3D. Image quality would be better with intracranial electrode mats or depth electrodes that are already implanted in people with severe epilepsy who are being evaluated for epilepsy surgery. For both electrode types, the new 3D information will enable better diagnosis and so targeting of drug treatment. It could also pave the way to suppression of seizures by deep brain electrical stimulation which could transform management in severe intractable epilepsy.It can offer the same benefits in imaging in epilepsy in neonates and infants.

Patients diagnosed with epilepsy will be asked to participate in the epilepsy EIT study, then up to 32 electrodes will be applied on the subjects' scalp or the EIT systems will be linked to the existing EEG video recording systems and EIT will be recorded at the same time using some or all of the available intracranial electrodes. It may also use some scalp EEG electrode placed on the scalp for clinical or research purposes. Following completion of the recording, scalp electrodes and any paste will be removed, the EIT system will be disconnected from the videoEEG. Collected data will be analysed and compared to other imaging data.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with epilepsy with either active seizures or interictal EEG changes (for scalp electrodes group)
* Any patient with epilepsy with either active seizures under evaluation for epilepsy surgery (for intracranial electrodes group)
* Ability to give informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Epilepsy patients recruited from the patients of National Hospital for Neurology and Neurosurgery in London.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
EIT images accuracy | three years

CONTACTS AND LOCATIONS:
Overall Officials: David S Holder, Professor, Principal Investigator — University College London, University College Hospital
Locations (1):
- EEG telemetry unit Neurophysiology National Hospital for Neurology and Neurosurgery, London, United Kingdom